CLINICAL TRIAL: NCT02794961
Title: Application of Humanized Anti-CD22 Antibody in CAR-T Therapy of B Cell Hematological Malignancies
Brief Title: CD22 Targeting CAR-T Therapy Against B Cell Hematological Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kai Lin Xu; Jun Nian Zheng (Other)
Collaborators: iCarTAB BioMed Inc. (Unknown)
Responsible Party: Sponsor-Investigator, Kai Lin Xu; Jun Nian Zheng, President, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AF-08/04.2
Record Dates: First submitted 2016-06-06; First posted 2016-06-09 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Recurrent or Refractory B Cell Malignancy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD22 CAR-T (Experimental): Enrolled patients will receive three escalating doses of autologous CAR-T.
  Interventions: Biological: CD22 CAR-T

INTERVENTIONS:
Biological: CD22 CAR-T — Autologous CAR-T cells with average 1*10^6 cells/kg body weight

SUMMARY:
CD19 expression on B cell frequently lost after CD19-targeting CAR-T therapy. In present study, we construct a CD22-targeting chimeric antigen receptor to overcome this issue.

DETAILED DESCRIPTION:
CD19 is an ideal target with great potential for treating B-cell-derived hematological malignancies. Although the complete remission rate is as high as 93% by using CD19-targeting CAR-T technology, approximately 60% patients will have recurrent disease. Among all the recurrent patients, two thirds is revealed to loss their CD19 expression on B cell surface. For overcoming this issue, we establish a new chimeric antigen receptor containing humanized single chain antibody sequence to target CD22 molecule on B cells.

ELIGIBILITY:
Inclusion Criteria:

* Greater than four years of age
* Survival time>12 weeks
* B cell hematological malignancies by pathological examination
* Chemotherapy failure or recurrent B cell malignancy
* Creatinine< 2.5mg/dl
* Glutamic-pyruvic transaminase, glutamic oxalacetic transaminase< 3 fold of normal level
* Bilirubin<2.0mg/dl
* Karnofsky Performance Status>50% at the time of screening
* Adequate pulmonary, renal, hepatic, and cardiac function
* Fail in autologous or allogenic haemopoietic stem cell transplantation
* Free of leukocytes removal contraindications
* Voluntarily join CAR-T clinical trial
* Understand and sign written informed consent

Exclusion Criteria:

* Pregnant or nursing women
* Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
* Feasibility assessment proves that the efficiency of transduction of lymphocyte is below 10% or the lymphocyte cannot be propagated.
* Abnormal vital signs
* Highly allergic constitution or history of severe allergies, especially allergy to interleukin-2
* General infection or local severe infection, or other infection that is not controlled
* Dysfunction in lung, heart, kidney and brain
* Severe autoimmune diseases
* Other symptoms that are not applicable for CAR-T

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | 12 months
  The B cells in peripheral blood of all enrolled patients will be monitored every week

CONTACTS AND LOCATIONS:
Overall Officials: KaiLin Xu, MD. Ph.D., Principal Investigator — Xuzhou Medical University
Locations (1):
- Affiliated hospital of Xuzhou medical college, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Haso W, Lee DW, Shah NN, Stetler-Stevenson M, Yuan CM, Pastan IH, Dimitrov DS, Morgan RA, FitzGerald DJ, Barrett DM, Wayne AS, Mackall CL, Orentas RJ. Anti-CD22-chimeric antigen receptors targeting B-cell precursor acute lymphoblastic leukemia. Blood. 2013 Feb 14;121(7):1165-74. doi: 10.1182/blood-2012-06-438002. Epub 2012 Dec 14. PMID 23243285